CLINICAL TRIAL: NCT03347539
Title: Adolescent Uptake of Implants on a Mobile Health Unit
Brief Title: Implants on Mobile Health Unit
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB17-0233
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Nexplanon: This group is participants who choose to receive the nexplanon implant. This group will only have one study interaction in the form of filling out a survey, at the time of implant.
  Interventions: Device: Nexplaon
- Removal participants: This group is participants who choose to remove the nexplanon implant. This group will only have one study interaction in the form of filling out a survey, at the time of removal. Anyone with a Nexplanon implant can have the implant removed on the mobile health unit and become part of this group - removal participants do not need to be in the Nexplanon group.

INTERVENTIONS:
Device: Nexplaon — This study is an exploratory study of user reasons for Nexplanon implant and removal, and NOT a study on the efficacy or safety of Nexplanon. Nexplanon has already been FDA approved and its efficacy and safety studied.
  Groups: Nexplanon

SUMMARY:
This study explores reasons why adolescents choose to receive a nexplanon implant and remove a Nexplanon implant. Nexplanon is provided as part of the standard of care on the University of Chicago mobile health unit. This study explores reasons for implantation and removal of Nexplanon on this mobile health unit.

ELIGIBILITY:
Inclusion Criteria:

* Be biologically female
* Be seeking reproductive healthcare on a mobile health unit
* Be interested in receiving Nexplanon for birth control.
* Be between 14 and 19 years of age.

Exclusion Criteria:

* Be biologically male
* Be 13 and younger or 20 and older.

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will be adolescent females seeking reproductive healthcare on a mobile health unit.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Reasons for choosing Nexplanon | One time, immediately before receiving implant.
  Information will be collected through a survey regarding why adolescents choose to receive Nexplanon.

SECONDARY OUTCOMES:
Reasons for choosing to remove Nexplanon | One time, immediately before removing implant.
  Information will be collected through a survey regarding why adolescents choose to remove Nexplanon.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Information regarding reasons for choosing the implant and choosing to remove will be shared with Merck, the maker of Nexplanon.
Supporting Information: CSR
Time Frame: Data will be shared after all data has been collected. This will be after December 2019. Data will be shared by analytical closeout date, in December 2021.